CLINICAL TRIAL: NCT04660149
Title: An Exploration Into the Young Patients' (< 50 Years) Expectations Following Primary Total Hip Arthroplasty: What Outcomes Are Important to Them? A Qualitative Study.
Brief Title: An Exploration Into the Young Patients' (< 50 Years) Expectations Following Primary Total Hip Arthroplasty
Acronym: YOUNG HIP
Status: Completed | Type: Observational
Sponsor: Bournemouth University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/IRAS/LM
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Total Hip Replacements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study seeks to explore between 6-7 patient participants' (18-50 years old inclusive) own expectations and hopes leading up to a THA, then to examine their own views on their recovery and rehabilitation post-operatively. A qualitative, longitudinal approach will be utilised for this research with a generic qualitative method analysing the verbal data taken during interviews with participants. A combination of semi-structured and narrative interview techniques will investigate the patients' individual expected outcomes and priorities for their recovery.

The study approach seeks to explore the patients' own views of a successful outcome of THA, it hopes to discover any potential themes of needs and priorities in the younger patient, and compare these to the standard way of measuring these outcomes by using PROMS. The outcome will contribute to determining what more can be done to improve the care currently in place for this increasing group of patients.

DETAILED DESCRIPTION:
To be confident that healthcare providers are providing the very best patient care in the instance of the younger patient it is essential to ask them their own interpretation of needs and priorities, and how they feel they can be met. There currently is an urgent need for further studies into the area of total hip arthroplasty in young patients, especially qualitative research defining the outcomes important to them after surgery. The considerably larger, older patient population undergoing this surgery often influence the way post-operative outcomes are measured (Larsson et al 2019, Mannion et al 2009, Wright and Young 1997, Wright et al 2000).

The study aims to discover and explore the following questions:

Are the priorities of the younger patient (< 50) being addressed and fulfilled when undergoing a THR? Are the current Outcome Measures identifying the priorities and required outcomes of the younger patient (< 50) undergoing a THR? The study will use a qualitative approach and method. Interviews will be conducted either face to face, via telephone or video calls dependent on participant preference. Semi-structured and narrative methods will be combined to encourage the participant to talk freely in regard to their own views and opinions on their surgery. Participants will also be asked to complete the Hip Disability and Osteoarthritis Hip Score (HOOS) at baseline (pre surgery), 6 weeks post-surgery and 6 months post-surgery time points to examine if this outcome measure illustrates a similar state to that which they described during their interviews.

With the participants' consent, these interviews will be recorded and transcribed by the Chief Investigator.

Participants will be assigned a study number on recruitment. All data will be anonymised and labelled with the appropriate participant's study number.

Audio recordings of qualitative interviews will be transcribed by the Chief Investigator and anonymised transcriptions will be stored on secure servers at Milton Keynes University Hospital (MKUH). The audio recordings will be deleted at the end of the study.

Consent forms, any paper case report forms (CRF) and completed HOOS will be filed in the site file which will be held in a secure, locked filing cabinet within the Research and Development Department at Milton Keynes University Hospital. Identifiable data will be kept separately from the outcome data (both paper and electronic).

No identifiable information will be shared with other persons at any point. The study plans to interview the participants at three different time points in their surgical journey. The first will be pre surgery (baseline) at around the time that the operative treatment is decided upon and the Surgeon has listed them for surgery. The second interview will be conducted around six weeks post operatively (+ 14 days), this will explore the patients' thoughts on their immediate post-operative recovery and how they feel they are progressing. The final time will be six months post-surgery (+ 30 days); this interview will examine the patients' own opinions on their surgical outcomes and their own interpretation of the success of the procedure. The HOOS will also be completed at each time point.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-50 years of age inclusive.
* Scheduled to undergo a primary THR in the index hip in the next 12-18 months. (Patients will still be eligible despite previously having a THR in the opposing hip)
* Able to provide informed consent.
* Ability to understand and communicate in English.

Exclusion Criteria:

* Under 18 years of age
* Over 50 years of age
* Undergoing a revision of THR in the index hip.
* Unable to provide informed consent or participate in study interviews.
* Unable or unwilling to complete follow up interviews.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients attending Milton Keynes University Hospital and scheduled to undergo a Primary Total hip replacement
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-04-11 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Are the priorities of the younger patient (< 50) being addressed and fulfilled when undergoing a THR? | 12-18 months
  The priorities and goals of the participant will be explored through the study interviews, these findings will be compared with the outcomes recorded when caring for these patients.
Are the current Outcome Measures identifying the priorities and required outcomes of the younger patient (< 50) undergoing a THR? | 12-18 months
  The data recorded in the interview will be compared with the Patient Reported Outcome Measures reported at the same time, to compare the two findings.

CONTACTS AND LOCATIONS:
Overall Officials: Louise Mew, Study Director — Research Nurse
Locations (1):
- Milton Keynes University Hospital, Milton Keynes, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No identifiable patient information is to be shared with any other researcher

REFERENCES:
- [Background] Larsson A, Rolfson O, Karrholm J. Evaluation of Forgotten Joint Score in total hip arthroplasty with Oxford Hip Score as reference standard. Acta Orthop. 2019 Jun;90(3):253-257. doi: 10.1080/17453674.2019.1599252. Epub 2019 Apr 1. PMID 30931686
- [Background] Mannion AF, Kampfen S, Munzinger U, Kramers-de Quervain I. The role of patient expectations in predicting outcome after total knee arthroplasty. Arthritis Res Ther. 2009;11(5):R139. doi: 10.1186/ar2811. Epub 2009 Sep 21. PMID 19772556
- [Background] Wright JG, Young NL. The patient-specific index: asking patients what they want. J Bone Joint Surg Am. 1997 Jul;79(7):974-83. doi: 10.2106/00004623-199707000-00003. PMID 9234873
- [Background] Wright JG, Young NL, Waddell JP. The reliability and validity of the self-reported patient-specific index for total hip arthroplasty. J Bone Joint Surg Am. 2000 Jun;82(6):829-37. doi: 10.2106/00004623-200006000-00009. PMID 10859102